CLINICAL TRIAL: NCT03567889
Title: An Open-Label, Randomized, Controlled Multi-Center Study of The Efficacy of Daromun (L19IL2 + L19TNF) Neoadjuvant Intratumoral Treatment Followed by Surgery and Adjuvant Therapy Versus Surgery and Adjuvant Therapy in Clinical Stage IIIB/C/D Melanoma Patients
Brief Title: Efficacy of Daromun Neoadjuvant Intratumoral Treatment in Clinical Stage IIIB/C/D Melanoma Patients
Acronym: NeoDREAM
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Philogen S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PH-L19IL2TNF-01/18; 2023-507119-36-00 (EU CTIS Number)
Record Dates: First submitted 2018-05-18; First posted 2018-06-26 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Melanoma Stage IIIB; Melanoma Stage IIIC; Melanoma Stage IIID
Keywords: Melanoma Stage IIIB; Melanoma Stage IIIC; Melanoma Stage IIID
MeSH Terms: conditions — Melanoma | interventions — daromun; Surgical Procedures, Operative; Chemotherapy, Adjuvant

STUDY DESIGN:
Intervention Model Description: Total patients: approximately 186. Daromun plus surgery and adjuvant therapy treatment group (Arm 1): 93 evaluable patients. Surgery and adjuvant therapy (Arm 2): 93 evaluable patients. Patients enrolled will be randomized to the two different arms of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Daromun plus Surgery and Adjuvant therapy (Experimental): Arm-1 patients will follow these steps:
  1. screening period,
  2. 4-week open-label treatment period,
  3. surgery within a maximum of 4 weeks,
  4. adjuvant therapy.
  Interventions: Drug: Daromun; Procedure: Surgery; Drug: Adjuvant therapy
- Surgery and adjuvant therapy (Active Comparator): Arm-2 patients will follow these steps:
  1. Screening period,
  2. direct surgery within 4 weeks from randomization,
  3. adjuvant therapy.
  Interventions: Procedure: Surgery; Drug: Adjuvant therapy

INTERVENTIONS:
Drug: Daromun — Patients will receive intratumoral administrations into injectable cutaneous, subcutaneous, and nodal tumors of Daromun once weekly for up to 4 weeks.
  Arms: Daromun plus Surgery and Adjuvant therapy
Procedure: Surgery — Patients will receive surgery.
Drug: Adjuvant therapy — Patients will receive adjuvant therapy at the investigator's discretion following the surgery.

SUMMARY:
The trial aims to evaluate the efficacy of Daromun neoadjuvant treatment followed by surgery and adjuvant therapy to improve in a statistically significant manner the recurrence-free survival (RFS) of Stage IIIB/C/D melanoma patients with respect to the standard of care (surgery and adjuvant therapy).

DETAILED DESCRIPTION:
The present study is an open-label, randomized, controlled, two-arm multi-center study of the efficacy of Daromun neoadjuvant intratumoral treatment followed by surgery and adjuvant therapy versus surgery and adjuvant therapy in clinical stage III B/C/D melanoma patients. 186 patients will be randomized in a 1:1 ratio to receive Daromun treatment followed by surgery and adjuvant therapy (Arm 1) or surgery and adjuvant therapy (Arm 2).

In both arms, follow-up for assessing recurrence-free survival will be performed up to five years after randomization. Survival information will also be collected in the following year (up to six years in total after randomization).

This is an open-label study, so there is no blinding.

Patients who successfully complete the screening evaluations and are eligible for participation in the study will be enrolled and randomly assigned (1:1) to two parallel treatment arms: Daromun plus surgery and adjuvant therapy (Arm 1) or surgery and adjuvant therapy (Arm 2).

To ensure a balance across treatment groups, stratified randomization with permuted block will be used and separate randomization list for each subgroup (stratum) will be produced. Patients will be stratified on the basis of the following prognostic factors:

* Stage of disease (3 levels): Stage IIIB vs. Stage IIIC vs Stage IIID
* Planned post-surgical adjuvant therapy (2 levels): anti-PD-1 and other adjuvant therapies.

The primary objective of the study is to demonstrate that a neoadjuvant Daromun treatment followed by surgery and adjuvant therapy improves in a statistically significant manner the recurrence-free survival (RFS) of Stage IIIB/C/D melanoma patients with respect to the standard of care (surgery and adjuvant therapy).

Primary endpoint of the study is RFS in a time-to-event analysis in the Daromun plus surgery and adjuvant therapy treatment group (Arm 1) versus the surgery plus adjuvant therapy control group (Arm 2). Analysis will be based on the "Intention To Treat" population.

The key secondary objective of the study is to demonstrate that a neoadjuvant Daromun treatment followed by surgery and adjuvant therapy improves in a statistically significant manner the overall survival (OS) of patients with resectable Stage IIIB/C/D melanoma patients with respect to the standard of care (surgery and adjuvant therapy).

For patients enrolled in both arms, local approved post-surgery adjuvant therapies (as part of the standard of care) are allowed and decided at the investigator's discretion. These include high-dose interferon- α2b, anti-CTLA-4 antibodies (e.g. Ipilimumab), anti-PD1 antibodies (e.g. Nivolumab, Pembrolizumab), targeted therapies (e.g. Dabrafenib + Trametinib), or other new local approved treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed diagnosis of clinical stage IIIB, IIIC, and IIID (AJCC 8th edition) locoregional melanoma that is eligible for complete surgical resection of all metastases (surgically resectable).
2. Eligible subjects must have measurable disease and must be candidate for intralesional therapy with at least one injectable cutaneous, subcutaneous, or nodal melanoma lesion (≥ 10 mm in longest diameter) or with multiple injectable lesions that in aggregate have a longest diameter of ≥ 10 mm.
3. Prior anti-tumor treatment for the primary melanoma lesion, including surgery and approved adjuvant treatments (e.g., radiotherapy, immune checkpoint inhibitors, BRAF/MEK inhibitors, etc.) is allowed. Before enrollment in the study, a wash-out period of 6 weeks is required and toxicities from prior treatments should be resumed to Grade ≤1.
4. Males or females, age ≥ 18 years.
5. ECOG Performance Status/WHO Performance Status ≤ 1.
6. Life expectancy of > 24 months.
7. Absolute neutrophil count > 1.5 x 109/L.
8. Hemoglobin > 9.0 g/dL.
9. Platelets > 100 x 109/L.
10. Total bilirubin ≤ 30 μmol/L (or ≤ 2.0 mg/dl).
11. ALT and AST ≤ 2.5 x the upper limit of normal (ULN).
12. Serum creatinine < 1.5 x ULN.
13. LDH serum level ≤ 1.5 x ULN.
14. Documented negative test for HIV, HBV and HCV. For HBV serology, the determination of HBsAg and anti-HBcAg Ab is required. In patients with serology documenting previous exposure to HBV (i.e. positive anti-HBsAg with not vaccination and/or positive anti-HBcAg Ab), negative serum HBV-DNA is also required.
15. All acute toxic effects (excluding alopecia) of any prior therapy must have resolved to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) (v4.03) Grade ≤ 1 unless otherwise specified above.
16. All women of childbearing potential (WOCBP) must have negative pregnancy test results at the screening. WOCBP must be using, from the screening to three months following the last study drug administration, highly effective contraception methods. WOCBP and effective contraception methods are defined by the "Recommendations for contraception and pregnancy testing in clinical trials" issued by the Head of Medicine Agencies' Clinical Trial Facilitation Group and which include, for instance, progesterone-only or combined (estrogen- and progesterone-containing) hormonal contraception associated with inhibition of ovulation, intrauterine devices, intrauterine hormone-releasing systems, bilateral tubal occlusion, vasectomized partner or sexual abstinence. Pregnancy test will be repeated at the safety visit (only WOCBP and only for patients in Arm 1).
17. Male patients with WOCBP partners must agree to use simultaneously two acceptable methods of contraception (i.e. spermicidal gel plus condom) from the screening to three months following the last study drug administration.
18. Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study.
19. Willingness and ability to comply with the scheduled visits, treatment plan, laboratory tests and other study procedures.

Exclusion Criteria

1. Uveal melanoma or mucosal melanoma
2. Evidence of distant metastases at screening.
3. Previous or concurrent cancer that is distinct in primary site or histology from the cancer being evaluated in this study except: cervical carcinoma in situ, curatively treated basal cell carcinoma, superficial bladder tumors (Ta, Tis & T1), second primary melanoma in situ or any cancer curatively treated ≥ 5 years prior to study entry.
4. Presence of active infections (e.g. requiring antimicrobial therapy) or other severe concurrent disease, which, in the opinion of the investigator, would place the patient at undue risk or interfere with the study.
5. History within the last year of acute or subacute coronary syndromes including myocardial infarction, unstable or severe stable angina pectoris.
6. Inadequately controlled cardiac arrhythmias including atrial fibrillation.
7. Heart insufficiency (> Grade II, New York Heart Association (NYHA) criteria).
8. LVEF ≤ 50% and/or abnormalities observed during baseline ECG and Echocardiogram investigations that are considered as clinically significant by the investigator.
9. Uncontrolled hypertension.
10. Ischemic peripheral vascular disease (Grade IIb-IV).
11. Severe diabetic retinopathy.
12. Active autoimmune disease.
13. History of organ allograft or stem cell transplantation.
14. Recovery from major trauma including surgery within 4 weeks prior to enrollment.
15. Known history of allergy to IL2, TNF, or other human proteins/peptides/antibodies or any other constituent of the product.
16. Breast feeding female.
17. Anti-tumor therapy (except small surgery) within 4 weeks before enrollment.
18. Previous in vivo exposure to monoclonal antibodies for biological therapy in the 6 weeks before enrollment.
19. Planned administration of growth factors or immunomodulatory agents within 7 days before enrollment.
20. Patient requiring or taking corticosteroids or other immunosuppressant drugs on a long-term basis will be evaluated case by case with the Sponsor for inclusion/exclusion in the study. Limited use of corticosteroids to treat or prevent acute hypersensitivity reactions is not considered an exclusion criteria.
21. Any conditions that in the opinion of the investigator could hamper compliance with the study protocol.
22. Previous enrolment and randomization in the same study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Estimated)
Dates: Start 2018-09-20 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Recurrence Free Survival (RFS) | From date of randomization until the date of the first recurrence or date of death from any cause, whichever occurs first assessed up to 60 months.
  Recurrence Free Survival (RFS) in a time-to-event analysis in the Daromun plus surgery and adjuvant therapy treatment group (Arm 1) versus the surgery and adjuvant therapy control group (Arm 2). Analysis will be performed for the "Intention To Treat" population.

SECONDARY OUTCOMES:
Overall survival (OS) | From date of randomization until the date of the first recurrence or date of death from any cause, whichever occurs first, assessed up to 72 months.
  Overall survival (OS) in the Daromun plus surgery and adjuvant therapy treatment group (Arm 1) versus surgery and adjuvant therapy (Arm 2), which will be evaluated in time to event analysis as key secondary endpoint.
Recurrence free survival (RFS) as determined by the local investigator | From date of randomization until the date of the first recurrence or date of death from any cause, whichever occurs first assessed up to 60 months.
  A sensitivity analysis to assess ascertainment bias will be performed on recurrence free survival. For this analysis the primary analysis definition of recurrence will be split into its two components and each will be analyzed separately. The first component/definition will be based on the unblinded assessment performed at the site - any new lesion detected by clinical evaluation which is confirmed by histopathology (biopsy or surgical specimen) and the second component/definition will be based on the assessment of a new lesion detected by allowed imaging modalities in a Blinded Independent Central Review and confirmed, wherever possible, by histological analysis. Each of these components will be analyzed separately using the same statistical model as the primary endpoint. Results from the two component analyses will be compared.
Event-free survival (EFS) | From date of randomization until the date of the first event as described above, assessed up to 60 months
  Event-free survival (EFS) defined as time from randomization to melanoma progression (irresectable stage III or stage IV disease), melanoma recurrence, treatment-related toxicity precluding surgery, treatment-related death, or melanoma-related death, whichever occurs first.
Adverse Events (AE) | From the inclusion in the study (signature of the informed consent form - ICF) until the first follow-up visit (up to approximately 5 months).
  Percentage of Patients in Each Treatment Group with AEs, AEs with CTCAE grade ≥3
Immune-related Adverse Events (irAEs) | From the inclusion in the study (signature of the informed consent form - ICF) until the end of follow-up (up to approximately 60 months).
  Occurrence of immune-related Adverse Events (irAEs)
Drug-Induced Liver Injury (DILI) | From the inclusion in the study (signature of the informed consent form - ICF) until the end of follow-up (up to approximately 60 months).
  Number of patients with Drug-Induced Liver Injury (DILI)
Adverse Events of Special Interest (AESI) | From the inclusion in the study (signature of the informed consent form - ICF) until the end of follow-up (up to approximately 60 months).
  Number of patients with Adverse Events of Special Interest (AESI)
Haematological/chemical Laboratory Abnormalities | From the inclusion in the study (signature of the informed consent form - ICF) until the end of follow-up (up to approximately 60 months).
  Percentage of Subjects with Haematological/chemical Laboratory Abnormalities
Electrocardiogram (ECG) and echocardiogram (ECHO) abnormalities | 1) day 0-14 (screening) for both arm; 2) at week 5 (Safety assessment) only for arm 1.
  Percentage of participants with Electrocardiogram (ECG) and echocardiogram (ECHO) abnormality findings. Data about QT/QTc intervals will be collected and analysed for QT/QTc prolongation potentially caused by treatment.
Physical examination | From the inclusion in the study (signature of the informed consent form - ICF) until the end of follow-up (up to approximately 60 months)
  Number of subjects with a clinically significant change from baseline in physical examination
Concomitant medication | From the inclusion in the study (signature of the informed consent form - ICF) until the end of follow-up (up to approximately 60 months)
  Number of subject with concomitant medication
Human anti-fusion protein antibodies (HAFA) | 1) day 0-14 (screening) for arm 1; 2) at week 5 (Safety assessment) for Arm 1; 3) at week 12 (only first follow-up) for Arm 1.
  Assessment of the formation of human anti-fusion protein antibodies (HAFA) against L19IL2 and L19TNF
Vital signs (blood pressure) | From the inclusion in the study (signature of the informed consent form - ICF) until the end of follow-up (up to approximately 60 months).
  Number of subjects with a clinically significant change from baseline in vital signs (blood pressure) by visit
Vital signals (heart rate) | From the inclusion in the study (signature of the informed consent form - ICF) until the end of follow-up (up to approximately 60 months)
  Number of subjects with a clinically significant change from baseline in vital signs (heart rate) by visit
Vital signals (body temperature) | From the inclusion in the study (signature of the informed consent form - ICF) until the end of follow-up (up to approximately 60 months)
  Number of subjects with a clinically significant change from baseline in vital signs (body temperature) by visit
Pathological responses | Assessed at the time of surgical resection of the tumor lesions.
  Pathological responses (categorized into pCR, near-pCR, pPR, pNR, according to INMC criteria) assessed at time of surgical resection.

OTHER OUTCOMES:
Local recurrence-free survival (LRFS) and distant metastasis-free survival (DMFS) | From date of randomization until the date of the first recurrence or date of death from any cause, whichever occurs first assessed up to 60 months
  Local recurrence-free survival (LRFS) and distant metastasis-free survival (DMFS) after randomization in the Daromun plus surgery and adjuvant therapy treatment group (Arm 1) versus surgery adjuvant therapy (Arm 2). LRFS is defined as survival free of loco-regional recurrence occurring at any time before systemic recurrence and other events are censored. DMFS is defined as survival free of systemic recurrence, including: 1) systemic recurrence outside the locoregional area at any time before or after locoregional relapse, 2) systemic recurrence with or without loco-regional relapse, or 3) death from cancer with no information on systemic recurrence.

CONTACTS AND LOCATIONS:
Locations (37):
- United States (19):
  - Mayo Clinic Hospital, Phoenix, Arizona
  - UC San Diego Moores Cancer Center, La Jolla, California
  - UC Irvine Health-Chao Family Comprehensive Cancer Center, Orange, California
  - Moffitt Cancer Center, Tampa, Florida
  - Winship Cancer Institute, Emory university, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Mayo Clinic, Rochester, Minnesota
  - Rutgers Cancer Institute, 195 Little Albany Street, New Brunswick, New Jersey
  - Ambulatory Care Center at NYC Langarone Health, New York, New York
  - Memorial Sloan Kettering Cancer Center - Main Campus, Ney York, New York
  - Duke University Medical Center - Duke Cancer Center, Durham, North Carolina
  - Ohio State University Wexner Medical Center, Columbus, Ohio
  - St. Luke's Cancer Center, Clinical Trial, 3rd floor, 1600 St. Luke's Blvd., Easton, Pennsylvania
  - Penn State Cancer Institute, Hershey, Pennsylvania
  - Fox Chase Cancer Center 333 Cottman Avenue, Philadelphia, Pennsylvania
  - The University of Texas M.D. Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute, University of Utah 2000 Circle of Hope, Salt Lake City, UT, Utah
  - VCU - McGlothlin Medical Education Center, Richmond, Virginia
- Spain (12):
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona
  - Fir Huvh Fundacio Institut De Recerca Hospital Universitari Vall De Hebron, Barcelona, Barcelona
  - Hospital Clinic Barcelona, Barcelona, Barcelona
  - El Hospital Universitario De Gran Canaria Dr. Negrin, Las Palmas de Gran Canaria, Canarie
  - Fundacion Onkologikoa Fundazioa, Donostia / San Sebastian, Gipuzkoa
  - MD Anderson Cancer Center, Madrid, Madrid
  - Hospital Universitario 12 de Octubre, Madrid, Madrid
  - Hospital Universitario Regional de Málaga, Málaga, Malaga
  - Hospital Clínico Universitario Virgen de la Arrixaca, Murcia, Murcia
  - Hospital Universitario Virgen De La Macarena, Seville, Sevilla
  - Hospital General Universitario de Valencia, Valencia
- Switzerland (6):
  - Universitätsspital Basel, Basel, Basel
  - Istituto Oncologico della Svizzera Italiana, Bellinzona, Bellinzona
  - Insel Gruppe AG, Bern, Canton of Bern
  - Hôpitaux Universitaires de Genève, Geneva, Canton of Geneva
  - Kantonsspital St.Gallen, Sankt Gallen, Canton of St. Gallen
  - Universitätsspital Zürich (USZ), Zurich, Canton of Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gorry C, McCullagh L, O'Donnell H, Barrett S, Schmitz S, Barry M, Curtin K, Beausang E, Barry R, Coyne I. Neoadjuvant treatment for stage III and IV cutaneous melanoma. Cochrane Database Syst Rev. 2023 Jan 17;1(1):CD012974. doi: 10.1002/14651858.CD012974.pub2. PMID 36648215
- [Derived] Miura JT, Zager JS. Neo-DREAM study investigating Daromun for the treatment of clinical stage IIIB/C melanoma. Future Oncol. 2019 Nov;15(32):3665-3674. doi: 10.2217/fon-2019-0433. Epub 2019 Sep 20. PMID 31538818